CLINICAL TRIAL: NCT04415632
Title: Effects of an Iso-energetic Low Glycemic Index (GI) Diet on Liver Fat Accumulation and Gut Microbiota Composition in Patients With Non- Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Low GI Diet Effects on Non-Alcoholic Fatty Liver Disease
Acronym: LGI-NAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 19042; 262245 (Other: IRAS); 19/EM/0291 (Other: REC)
Record Dates: First submitted 2020-04-20; First posted 2020-06-04 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Fatty Liver; Nutritional and Metabolic Disease
MeSH Terms: conditions — Fatty Liver; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LGI Diet (Experimental): low glycemic index diet
  Interventions: Other: low glycemic index diet
- HGI Diet (Other): High glycemic index diet
  Interventions: Other: High glycemic index diet

INTERVENTIONS:
Other: low glycemic index diet — • Three-day cycle menu of LGI diet will be designed and supplied to each participant in an amount designed to meet their estimated energy requirements. The percentage energy from protein, fat and carbohydrate will be the same in the two diets. Each diet period of the trial will last for two weeks.
  Other Names: LGI
  Arms: LGI Diet
Other: High glycemic index diet — Three-day cycle menu of HGI diet will be designed and supplied to each participant in an amount designed to meet their estimated energy requirements. The percentage energy from protein, fat and carbohydrate will be the same in the two diets. Each diet period of the trial will last for two weeks.
  Other Names: HGI
  Arms: HGI Diet

SUMMARY:
A 2 x 2 cross-over dietary intervention trial designed to investigate the effects of low glycemic index (LGI) versus high glycemic index (HGI) diet on hepatic fat accumulation and gut microbiota composition in participants with NAFLD.

Participants will be allocated randomly to a 2-week either high GI (HGI) or low GI (LGI) diet followed by a 4-week wash-out period and then the LGI or HGI diet, opposite to the first 2-weeks (N= 16).

ELIGIBILITY:
Inclusion Criteria:

* • Adult males and females aged from 18 to 65 years (balanced number).

  * Detected NAFLD by CAP-FibroScan™ >288dB/m or by MRI-PDFF) > 5% fat of liver weight.
  * Body mass index ≥ 25 kg/m2
  * Have current moderate to high GI diet intake of ≥ 60 (Assessed from a completed 7-day food diary).
  * Abdominal obesity (Waist circumference > 102 cm for males and > 88 cm for females)
  * Able to give informed consent.
  * Able to undergo MRI/S and CAP-FibroScan™.

Exclusion Criteria:

* • Current smokers and excessive alcohol drinkers (> 14 units/week).

  * Perimenopausal (irregular periods) women.
  * Participants with other liver abnormalities.
  * Participants with history of gastrointestinal surgeries, depression, eating disorders or difficulties.
  * Participants using pharmacologic agents for obesity or NAFLD.
  * Participants with type 1 diabetes.
  * Participants with type 2 diabetes on second line medications (eg GLP-1 analogues, sulfonylureas).
  * Participation in any other trial in the last 3 months.
  * Participants on any special diets (e.g. vegetarians).
  * Intolerance to foods included in the diet plan.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
liver fat content | At baseline
  To assess the difference in liver fat content between LGI and HGI diet groups in participants with NAFLD using MRI/S
liver fat content | 2 weeks
  To assess the difference in liver fat content between LGI and HGI diet groups in participants with NAFLD using MRI/S

SECONDARY OUTCOMES:
Gut microbial composition | At baseline
  To assess the difference in gut microbiota composition between LGI and HGI diet groups in participants with NAFLD using 16S sequencing of rRNA
Gut microbial composition | 2 weeks
  To assess the difference in gut microbiota composition between LGI and HGI diet groups in participants with NAFLD using 16S sequencing of rRNA
Blood glucose level | At baseline
  To assess the differences in blood glucose levels between LGI and HGI diet groups in participants with NAFLD using Horiba automated analyser.
  .
Blood glucose level | 2 weeks
  To assess the differences in blood glucose levels between LGI and HGI diet groups in participants with NAFLD using Horiba automated analyser.
Blood insulin levels | At baseline
  To assess the differences in blood insulin levels between LGI and HGI diet groups in participants with NAFLD using radioimmunoassay methods .
Blood insulin levels | 2 weeks
  To assess the differences in blood insulin levels between LGI and HGI diet groups in participants with NAFLD using radioimmunoassay methods .
blood liver function tests | At baseline
  To assess the differences in liver function biomarkers between LGI and HGI diet groups in participants with NAFLD using Horiba automated analyser. The blood liver function tests (LFTs) to be assessed are GGT(Gamma-Glutamyl Transferase), ALP(Alkaline Phosphatase), AST(Aspartate Amino Transferase), and ALT(Alanine Amino Transferase)
blood liver function test | 2 weeks
  To assess the differences in liver function biomarkers between LGI and HGI diet groups in participants with NAFLD using Horiba automated analyser. The blood liver function tests (LFTs) to be assessed are GGT(Gamma-Glutamyl Transferase), ALP(Alkaline Phosphatase), AST(Aspartate Amino Transferase), and ALT(Alanine Amino Transferase)
blood lipids levels | At baseline
  To assess the differences in blood lipids levels between LGI and HGI diet groups in participants with NAFLD using Horiba automated analyser. The blood lipids biomarkers to be assessed are Total Cholesterol, Free Fatty Acids, High-density lipoprotein, low-density lipoprotein, Triglycerides.
blood lipids levels | 2 weeks
  To assess the differences in blood lipids levels between LGI and HGI diet groups in participants with NAFLD using Horiba automated analyser. The blood lipids biomarkers to be assessed are Total Cholesterol, Free Fatty Acids, High-density lipoprotein, low-density lipoprotein, Triglycerides.
blood gut hormones levels | At baseline
  To assess the differences in blood gut hormones levels between LGI and HGI diet groups in participants with NAFLD using radioimmunoassay (RIA) or Sandwich ELISA methods. The blood gut hormones to be assessed are Glucagon, Leptin, Ghrelin, PYY (Peptide YY), GLP-1 (Glucagon-like peptide 1).
blood gut hormones levels | 2 weeks
  To assess the differences in blood gut hormones levels between LGI and HGI diet groups in participants with NAFLD using radioimmunoassay (RIA) or Sandwich ELISA methods. The blood gut hormones to be assessed are Glucagon, Leptin, Ghrelin, PYY (Peptide YY), GLP-1 (Glucagon-like peptide 1).
Plasma Short Chain Fatty Acids (SCFAs) | At baseline
  To investigate the differences in plasma SCFAs between LGI and HGI diet groups in participants with NAFLD.
Plasma Short Chain Fatty Acids (SCFAs) | 2 weeks
  To investigate the differences in plasma SCFAs between LGI and HGI diet groups in participants with NAFLD.
Anthropometric measurements | At baseline
  Weight in kg, Height in meters will be combined to report BMI kg/m^2 or each study arm
Anthropometric measurements | 2 weeks
  Weight in kg, Height in meters will be combined to report BMI kg/m^2 or each study arm
Body composition Fat Mass | At baseline
  Bio-electrical Impedance analysis (BIA) will be used to assess the body composition of fat mass %.
Body composition Fat Mass | 2 weeks
  Bio-electrical Impedance analysis (BIA) will be used to assess the body composition of fat mass %.
Body composition Muscle Mass | At baseline
  Bio-electrical Impedance analysis (BIA) will be used to assess the body composition of muscle mass %.
Body composition Muscle Mass | 2 weeks
  Bio-electrical Impedance analysis (BIA) will be used to assess the body composition of muscle mass %.
Body composition Water Content | At baseline
  Bio-electrical Impedance analysis (BIA) will be used to assess the body composition of water content %.
Body composition Water Content | 2 weeks
  Bio-electrical Impedance analysis (BIA) will be used to assess the body composition of water content %.
Visual analogue scales (VAS) | through study completion, an average of two weeks
  Visual analogue scales (VAS) in 0 to 10 cm scale will be used to assess the participant's subjective appetite (hunger and fullness) during the each study arm.

CONTACTS AND LOCATIONS:
Locations (1):
- NIHR Nottingham Clinical Research Facility Nottingham Digestive Diseases Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Within a five-year timeframe, the final anonymized trial data will be uploaded to the https://rdmc.nottingham.ac.uk public repository after consistency and quality have been verified by the project team and publication of the results. Data from this trial are intended to be presented at local and international conferences including those attended by clinicians and dietitians and will also be used as part of a Philosophy Doctorate thesis. Publications will be in peer reviewed journals. No participant will be identified in any of these publications.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: within five years time-frame
Access Criteria: Public repository. presented at local and international conferences. part of a Philosophy Doctorate thesis
URL: https://rdmc.nottingham.ac.uk

REFERENCES:
- [Derived] Al-Awadi A, Grove J, Taylor M, Valdes A, Vijay A, Bawden S, Gowland P, Aithal G. Effects of an isoenergetic low Glycaemic Index (GI) diet on liver fat accumulation and gut microbiota composition in patients with non-alcoholic fatty liver disease (NAFLD): a study protocol of an efficacy mechanism evaluation. BMJ Open. 2021 Oct 7;11(10):e045802. doi: 10.1136/bmjopen-2020-045802. PMID 34620653